CLINICAL TRIAL: NCT00541294
Title: Diagnosis of Tuberculosis Infection in HIV Co-infected Children
Acronym: ThrasherIGRA
Status: Completed | Type: Observational
Sponsor: Case Western Reserve University (Other)
Collaborators: Thrasher Research Fund (Other)
Responsible Party: Principal Investigator, Anna Maria Mandalakas, Professor, Baylor College of Medicine
Other Study IDs: RES104272
Record Dates: First submitted 2007-10-05; First posted 2007-10-10 (Estimated); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: Latent Tuberculosis Infection; Tuberculosis; HIV Infections
Keywords: Tuberculosis; HIV; Diagnostics; Pediatrics
MeSH Terms: conditions — Latent Tuberculosis; Tuberculosis; HIV Infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- B: M.tb unexposed HIV-infected and uninfected children <15 years of age
- A: M.tb exposed HIV-infected and uninfected children <15 years of age

SUMMARY:
Background: The TB and HIV epidemics are closely linked in developing countries, where 450,000 children die from HIV annually. TB is a major cause of death in HIV-infected children and is reversing gains made in child survival.

The traditional tuberculin skin test (TST) has limited diagnostic accuracy for detecting TB infection. Adult studies suggest that new blood-based diagnostic TB testing offers a quicker, more accurate way to diagnose TB infection. Such diagnostic testing may directly guide clinical management and preventive strategies in immune-suppressed HIV-infected children, who are at high risk of becoming TB diseased following infection. Data regarding the usefulness of these tests in children is currently limited.

Objective(s) and Hypothesis(es): The investigators hypothesize that blood-based TB diagnostic testing can accurately identify children with TB infection. In a community with high rates of TB and HIV infection, the following specific aims will be investigated in HIV-infected and uninfected children:

1. assess the agreement between the TST and blood-based diagnostic testing,
2. compare the performance of the TST and blood-based diagnostic testing to a standardized history of TB exposure,
3. measure the impact of age, nutritional and immune status on children's response to blood-based testing,
4. describe factors that might modify children's response to testing over time, and 5) examine the effect of environmental exposures and previous vaccination on the TST, blood-based testing and other measures of immune responses to TB.

Potential Impact: The benefits of an accurate, rapid diagnostic test of TB infection in children include 1) timely institution of treatment for TB infection to prevent severe disease and mortality, and 2) preclusion of over diagnosis and treatment. Treatment of childhood TB infection also prevents future contagious adult disease, thus decreasing community transmission. Blood-based diagnostic testing may also be able to identify children that are more likely to become ill following TB infection. Therefore, blood-based diagnostic testing has great potential to improve TB control and the health of HIV-infected and uninfected children, their households and communities.

ELIGIBILITY:
Inclusion Criteria:

* age less than 15 years
* completion of informed consent

Exclusion Criteria:

* less than 3 months of age
* documented anemia
* recent diagnosis of tuberculosis
* receiving treatment for tuberculosis

Ages: 3 Months to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: HIV seropositive and seronegative South African children (6months to 15years) with and without M.tb exposure
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2008-01-15 (Actual); Primary Completion 2011-02-22 (Actual); Study Completion 2011-02-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anna M Mandalakas, MD, PhD, Principal Investigator — Baylor College of Medicine; Anneke C Hesseling, MD, MS, Principal Investigator — University of Stellenbosch
Locations (1):
- Despond TuTu TB Centre, Stellenbosch University, Tygerberg, Western Cape, South Africa